CLINICAL TRIAL: NCT03092908
Title: Mature Vinegar Prophylaxis Against Recurrent Calcium Oxalate Nephrolithiasis - a Prospective Randomized Controlled Trial
Brief Title: Mature Vinegar Prophylaxis Against Recurrent Calcium Oxalate Nephrolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MRER(62)2016
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Nephrolithiasis
Keywords: calcium oxalate; nephrolithiasis; Mature vinegar; prophylaxis
MeSH Terms: conditions — Nephrolithiasis | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Administer 5 ml placebo (purified water) three times a day.
  Interventions: Dietary Supplement: placebo (water)
- Intervention group (Experimental): Administer 5 ml mature vinegar (Brand: Ninghuafu) three times a day.
  Interventions: Dietary Supplement: mature vinegar

INTERVENTIONS:
Dietary Supplement: mature vinegar — Administer 5 ml mature vinegar (Brand: Ninghuafu) three times a day.
  Arms: Intervention group
Dietary Supplement: placebo (water) — Administer 5 ml placebo (water) three times a day.
  Arms: Control group

SUMMARY:
Kidney stones are one of the most common disorders of the urinary tract and cause a great deal of morbidity and economic loss. Because of the high recurrence rate, researchers are interested in finding medicinal therapies to prevent kidney stone recurrence. Vinegar is consumed worldwide as a food condiment and preservative. The mature vinegar, also called black vinegar, is an inky-black vinegar aged for a malty, woody, and smoky flavor. It is popular in the north of China as a dipping sauce, particularly for dumplings.

Some studies promote vinegar for its medicinal properties, as a tonic which may lower blood pressure and cholesterol level. Our national epidemiological data in China showed that consumed more mature vinegar was associated with decreased risk of kidney stones formations. Furthermore, our previous in vivo study found that mature vinegar could inhibit renal calcium oxalate crystals formation in rat model. These findings inspire us to clarify the nephrolithiasis prevention effect of mature vinegar in a clinical trial. In this study, investigators would like to examine the efficacy of mature vinegar prophylaxis for preventing recurrent calcium oxalate nephrolithiasis.

DETAILED DESCRIPTION:
Background: Kidney stones are one of the most common disorders of the urinary tract and cause a great deal of morbidity and economic loss. Because of the high recurrence rate, researchers are interested in finding medicinal therapies to prevent kidney stone recurrence. Vinegar is consumed worldwide as a food condiment and preservative. The mature vinegar, also called black vinegar, is an inky-black vinegar aged for a malty, woody, and smoky flavor. It is popular in the north of China as a dipping sauce, particularly for dumplings.

Some studies promote vinegar for its medicinal properties, as a tonic which may lower blood pressure and cholesterol level. Our national epidemiological data in China showed that consumed more mature vinegar was associated with decreased risk of kidney stones formations. Furthermore, our previous in vivo study found that mature vinegar could inhibit renal calcium oxalate crystals formation in rat model (unpublished). These findings inspire us to clarify the nephrolithiasis prevention effect of mature vinegar in a clinical trial. In this study, investigators would like to examine the efficacy of mature vinegar prophylaxis for preventing recurrent calcium oxalate nephrolithiasis.

Methods: A prospective randomized, controlled, single-center clinical trial will be performed at the First Affiliated Hospital of Guangzhou Medical University from March 2017 to March 2022.

Intervention: 80 subjects are randomly assigned in a 1:1 ratio to receive mature vinegar or placebo. The sequence of randomization is computer generated and are performed by the hospital's pharmacy service, whoever administer 5 ml mature vinegar (Brand: Ninghuafu) three times a day and placebo as liquid of the same type in identical bottles. The subjects, the attending urologist, and the investigators are not aware of study arm assignments until the final assessment of outcome.

From the beginning of invention, participants will be scheduled to receive a brief (< 10 min) individual telephone contact once per month and weekly text messages. The telephone contacts are conducted by intervention staff and followed a standard script. Text message are provided once per week and are used to remind participants in invention group of drinking mature vinegar.

Sample size estimation: According to non-continuous sample size calculation formula, , where P1 is 3-year stone recurrence rate in normal group , P2 is 3-year recurrence rate in mature vinegar group, P is (P1 + P2)/2. According to our preliminary clinical data, the 3-year stone recurrence rate in normal group between 30% and 50%. Assume P1 =40%. The vinegar invention would reduce the risk of recurrence by about three fourth. The 3-year stone recurrence rate after mature vinegar is 10% (P2). Using 95% confidence interval, an α error of 5%, and a power of 80%, the minimum sample size was estimated to be 32 subjects for each of the study groups. To account for subjects lost to follow-up and study withdrawals, this number is increased to 40.

Data collection and follow-up: Each subject's medical history is taken, a physical examination is performed, and the subject's weight, height, body mass index, blood pressure, education, income, employment status, smoking status, and alcohol consumption are measured and recorded. Assessment staff are masked to prior data at each assessment to minimize potential bias.

24-h urine and serum specimens are obtained at baseline (with values documented as the average of the two sets of measurements performed before randomization), 3 months after rafter randomization, half a year after randomization, and at yearly intervals during the 3 years of the study.

Outcome Measures: The primary outcome measure is the time to the first recurrence of a symptomatic renal stone or the presence of asymptomatic renal stone or the presence of a radiographically identified stone. In the event of a recurrence, the treatment is considered to have failed, and the patient will be withdrawn from the trial. If there are no recurrences, patients will be followed until the third annual visit (month 36). Patients who required treatment with thiazides or allopurinol for conditions such as hypertension or gout will be withdrawn from the trial.

Recurrences are considered to be either silent or symptomatic. Silent recurrences are diagnosed on the basis of renal ultrasound performed at 3 months, 6 months, 1 year, 2 year, 3 year after randomization. If renal stones are detected, CT will also be performed. The imaging studies will be performed by a central radiologic service, and the radiologist have no knowledge of the trial or the group assignment. A recurrence is classified as silent if a previously unreported stone was detected in the absence of symptom. A symptomatic recurrence is defined as typical renal colic, an episode hematuria, or the expulsion or removal of a previously undiscovered stone. If a symptomatic recurrence is documented on the basis of renal colic or hematuria, the recurrence will to be confirmed radiographically.

Secondary outcome measures include change in 24-h urine compositions (calcium excretion, oxalate excretion, etc.), serum calcium, phosphate, creatinine, and uric acid.

Statistical Analysis: The analysis is based on the intention-to-treat principle. Investigators use Kaplan-Meier analyses to determine the cumulative incidence of recurrent stones, and investigators use Cox proportional-hazards regression to determine the crude and adjust relative risks of recurrence.

For the analysis of the urinary indexes, investigators compare the two groups with respect to the absolute change from the base-line value at each time point. These comparisons are carried out with use of the Mann-Whitney test. Base-line continuous variables are compared with use of the Mann-Whitney test and Student's t-test whenever appropriate; categorical variables are compared with use of Fisher's exact test. A P value of less than 0.05 is considered to indicate statistical significance. All reported P values are two-side.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female > 18 years;
2. History of recurrent nephrolithiasis, with one or more calcium oxalate or mixed (calcium oxalate and phosphate, calcium oxalate and uric acid) stone formation over the last 5 years; the stone had been removed completely confirmed by CT scan;
3. No current treatment for the prevention of recurrent stones except for the advice to increase water intake;
4. Residence in the area of Guangzhou, China;
5. Written informed consent

Exclusion Criteria:

1. Obstructive uropathy, chronic urosepsis, renal failure (serum creatinine > 177 umol/L), renal tubular acidosis, primary hyperparathyroidism, primary hyperoxaluria, bowel resection, inflammatory bowel disease, pure uric acid and cystine stones, medullary sponge kidney;
2. Active peptic ulcer disease, gastric esophagus reflux; Past history of peptic ulcer disease;
3. Participants who had a known the vinegar effect for stone formation;
4. Concomitant clinical conditions that might affect completion of the study or jeopardize data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of renal stone | 3 years
  The first recurrence of a symptomatic renal stone or the presence of asymptomatic renal stone or the presence of a radiographically identified stone.

SECONDARY OUTCOMES:
24-h urine compositions | 3 years
  Change in 24-h urine compositions (calcium excretion, oxalate excretion, etc.)
serum calcium | 3 years
  Change in serum calcium
serum creatinine | 3 years
  Change in serum creatinine
serum uric acid | 3 years
  Change in serum uric acid

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China